CLINICAL TRIAL: NCT00139750
Title: A Double-Blind, Placebo-Controlled, Randomized, Multicenter Study Evaluating The Efficacy And Safety Of CP-526,555 In Smokers Motivated To Stop Smoking
Brief Title: 12 Week Evaluation of the Safety and Efficacy of 3 Doses of CP-526,555 and Placebo for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3051046
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2007-06-04 (Estimated); Status verified 2007-06

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

INTERVENTIONS:
Drug: CP-526,555 (varenicline)

SUMMARY:
The purpose of the study is to examine the safety and efficacy and dose-response relationship of three doses of CP-526,555 for 12 weeks compared with placebo for smoking cessation; including post-treatment follow-up of smoking status to one year from randomization. A small satellite protocol (A3051048) investigated safety of a second course of therapy in subjects who did not quit.

ELIGIBILITY:
Inclusion Criteria:

* Cigarette smokers who are motivated to stop smoking and have smoked an average of at least 10 cigarettes per day

Exclusion Criteria:

* Subjects who have used a nicotine replacement product within 30 days of the study screening visit or intend to use it during the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2004-12; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
4-week continuous quit rate (CQR) for Weeks 9-12

SECONDARY OUTCOMES:
Continuous abstinence for Weeks 9-52 and Weeks 9-24
Long-term quit rate at Week 52
4-week CQR for Weeks 4-7
7-day point prevalence of asbtinence Weeks 12, Week 24, and Week 52
Continuous abstinence from TQD (Week 1) through Week 12
Weekly average number of cigarettes smoked per day for Weeks 1-12
Evaluation of withdrawal symptoms by the Minnesota Nicotine Withdrawal Scale
Evaluation of smoking satisfaction by the Smoking Effects Inventory
Evaluation of urge to smoke by the Brief Questionnaire of Smoking Urges

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (15):
- Japan (15):
  - Pfizer Investigational Site, Noda, Chiba
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Ohita, Ohita
  - Pfizer Investigational Site, Beppu-shi, Oita Prefecture
  - Pfizer Investigational Site, Toyonaka, Osaka
  - Pfizer Investigational Site, Tosu, Saga-ken
  - Pfizer Investigational Site, Hamamatsu, Shizuoka
  - Pfizer Investigational Site, Edogawa-ku, Tokyo
  - Pfizer Investigational Site, Minato-ku, Tokyo
  - Pfizer Investigational Site, Musashino, Tokyo
  - Pfizer Investigational Site, Setagaya-ku, Tokyo
  - Pfizer Investigational Site, Shinagawa-ku, Tokyo
  - Pfizer Investigational Site, Toshima-ku, Tokyo

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Nakamura M, Oshima A, Ohkura M, Arteaga C, Suwa K. Predictors of lapse and relapse to smoking in successful quitters in a varenicline post hoc analysis in Japanese smokers. Clin Ther. 2014 Jun 1;36(6):918-27. doi: 10.1016/j.clinthera.2014.03.013. Epub 2014 May 5. PMID 24811751
- [Derived] Nakamura M, Oshima A, Fujimoto Y, Maruyama N, Ishibashi T, Reeves KR. Efficacy and tolerability of varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, in a 12-week, randomized, placebo-controlled, dose-response study with 40-week follow-up for smoking cessation in Japanese smokers. Clin Ther. 2007 Jun;29(6):1040-56. doi: 10.1016/j.clinthera.2007.06.012. PMID 17692720
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051046&StudyName=+12+Week+Evaluation+of+the+Safety+and+Efficacy+of+3+doses+of+CP%2D526%2C555+and+Placebo+for+Smoking+Cessation